CLINICAL TRIAL: NCT06126562
Title: A Phase I Clinical Study to Evaluate the Pharmacokinetic Profile and Safety of Lanifibranor After Single Dose and Multiple Doses in Healthy Adult Chinese Subjects
Brief Title: A Pharmacokinetic Study of Lanifibranor in Healthy Adult Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNLN-I-01
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Pharmacokinetic
MeSH Terms: interventions — lanifibranor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lanifibranor 800 mg (Experimental): In Part A, lanifibranor 800 mg is given as a single dose (followed by 14 days follow-up).
  In Part B, lanifibranor 800 mg is given once daily for 7 consecutive days (followed by 7 days follow-up).
  Interventions: Drug: Lanifibranor
- Lanifibranor 120 mg (Experimental): In Part A, lanifibranor 1200 mg is given as a single dose (followed by 14 days follow-up).
  In Part B, lanifibranor 1200 mg is given once daily for 7 consecutive days (followed by 7 days follow-up).
  Interventions: Drug: Lanifibranor

INTERVENTIONS:
Drug: Lanifibranor — Lanifibranor is a pan-peroxisome proliferator-activated receptor (PPAR) agonist.

SUMMARY:
This will be a randomized, open-label parallel design and single centre study conducted at the 1st hospital affiliated to Jilin University. Approximately 24 healthy Chinese volunteers, male and female will be recruited and divided into two equal groups (12 subjects per dose). The primary objective of this study is to evaluate the pharmacokinetic profile of lanifibranor after single dose and multiple doses 800 and 1200 mg in healthy adult Chinese subjects. The secondary objective is to evaluate the safety of lanifibranor after single dose and multiple doses 800 and 1200 mg in healthy adult Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years (both inclusive) at the time of signing the informed consent form (ICF), regardless of gender;
* Male subjects body weight ≥ 50 kg and female subjects body weight ≥ 45 kg, with a body mass index (BMI) of 18-28 kg/m2 (both inclusive);
* No clinically significant findings in medical history, physical examination, 12-lead ECG, vital signs, laboratory tests, etc.;
* Normal clinical laboratory test values at screening and baseline (Day 1) or judged as not clinically significant by the investigator and/or sponsor;
* Alanine aminotransferase ≤ 1.1 × upper limit of normal (ULN), aspartate aminotransferase ≤ 1.2 × ULN; normal renal function, estimated glomerular filtration rate (eGFR) > 60 mL/min/1.73 m2 at screening.
* Subjects need to understood the study, agree to voluntarily participate in the study, to comply with the study requirements, and provide written informed consent;
* Female subjects of childbearing potential must agree to use 2 highly effective methods of contraception, barrier contraception, during the study and within 30 days after one of which must be the study treatment. Female subjects must have a negative serum pregnancy test at screening and baseline (Day 1).
* Male subjects and their female partners of childbearing potential must agree to use 2 highly effective methods of contraception (as defined above), one of which must be a barrier method, during the study and for 90 days after receiving the study drug.

Exclusion Criteria:

* History or evidence of respiratory, circulatory, endocrine, urinary, digestive, immunological, reproductive, hematological, neurological, or psychiatric disorders, especially any history that may affect drug absorption, distribution, metabolism, and excretion.
* Subjects who are positive for any of the following: hepatitis B virus surface antigen (HBs-Ag), hepatitis C virus antibody (anti-HCV), human immunodeficiency virus antibody (anti-HIV), and treponema pallidum antibody (anti-TP).
* Subjects with any of the following conditions within 6 months prior to screening: Unstable body weight, Women with irregular menstruation or ovulation, including but not limited to women with Stein-Leventhal syndrome and perimenopausal women with abnormal ovulation, History of osteoporosis or fracture, History of oedema peripheral at any site, History of gallbladder disease, including but not limited to cholelithiasis, and cholecystitis, History of hypoglycemia or events highly suspicious of hypoglycaemia.
* Current tissue dysplasia or history of malignancy (including lymphoma and leukemia) within the past 5 years, except for successfully cured non-metastatic basal cell carcinoma or squamous cell carcinoma or localized cervical carcinoma in situ.
* Pregnant, lactating women, or women planning to become pregnant during the study or within 30 days of study drug administration.
* Treatment with another study drug or device within 3 months before study drug administration; or less than 5 half-lives from treatment with another study drug or device at screening, whichever is longer.
* Known hypersensitivity or intolerance to lanifibranor or any of the excipients, and allergic constitution.
* Consumption of more than 28 units of ethanol per week, or a history of alcohol abuse, at any time within 6 months prior to study drug administration.
* Smoking more than 5 cigarettes per day or consuming an equivalent amount of nicotine or nicotine-containing products within 6 months before screening, or an inability to discontinue the use of any tobacco products during the study.
* Taking prescription drugs (excluding oral and other contraceptives [e.g., long-acting formulations, transdermal contraceptives, and intrauterine devices]), including nonsteroidal anti-inflammatory drugs, sucralfate, drugs known to decrease metabolism or increase bioavailability, traditional Chinese medicine preparations, melatonin, or other nutritional supplements, within 14 days or 5 half-lives (whichever is longer) before study drug administration, or taking over-the-counter drugs, vitamins, or supplements (including cod-liver oil) within 7 days before study drug administration.
* Consuming products containing alcohol, caffeine, or xanthines, Seville oranges, and grapefruit or grapefruit juice within 72 hours prior to study drug administration.
* Engagement in strenuous activity (e.g., exercise) within 96 h (4 days) before admission to the clinical research unit (CRU) and throughout the study.
* Donation of more than 500 mL of blood or significant blood loss within 90 days prior to admission to the CRU.
* History or evidence of poor venous access or hemorrhagic disorder.
* History of drug use, drug abuse, or positive urine drug test.
* Any condition that, as determined by the investigator, may pose a safety risk to the subject during the study or may interfere with the study's conduct, or the investigator believes that the subject may not be able to complete the study or comply with its requirements.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  Maximum plasma drug concentration
Area under the plasma concentration-time curve | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  The area enclosed by the blood concentration curve to the timeline
Time to maximum concentration (Tmax) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  The time required to reach peak concentration after administration
Apparent volume of distribution (Vd/F) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  Drug dose reach a dynamic balance in the body the body and blood drug concentration ratio constant
Apparent plasma clearance (CL/F) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  The volume of plasma with drug cleared per unit of time
Plasma elimination half-life (t1/2) | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  The time it takes for the terminal phase blood concentration to drop by half
Time to maximum concentration at steady state (Tmax, ss) in Part B | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  The time required to reach peak steady-state concentration after administration
Maximum concentration at steady state (Cmax, ss) in Part B | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  The maximum blood drug concentration that occurs after stabilization
Minimum concentration at steady state (Cmin, ss) in Part B | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  The minimum blood drug concentration that occurs after stabilization
Average steady-state plasma concentration (Cav, ss) in Part B | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  The plasma concentration at which the rate of administration and rate of elimination are in equilibrium.

SECONDARY OUTCOMES:
Adverse event rate | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  The occurrence rate of all adverse events (AEs), and adverse events of special interest (AESI) and serious adverse events (SAEs).
Adverse event rate | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, 120, 168 hours after dose.
  The occurrence rate of abnormal clinical laboratory tests, vital signs, physical examination and 12 lead-electrocardiogram (ECG).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China